CLINICAL TRIAL: NCT02268474
Title: Prospective, Randomized, Controlled Split-Face Study of the Excel V 532nm KTP Laser for the Treatment of Erythematotelangiectatic Rosacea and Papulopustular Rosacea
Brief Title: Excel V 532 nm KTP Laser for Treatment of Erythematotelangiectatic Rosacea & Papulopustular Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-14-EV04
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Erythematotelangiectatic Rosacea; Papulopustular Rosacea
Keywords: 532nm; Excel V; Cutera; Laser; Laser Light; PDL; 595nm; Flash Lamp
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 532nm KTP Laser vs 595nm Pulse Dye Laser (Experimental): This is a single-center prospective, randomized, controlled split-face study in 20 subjects diagnosed with Erythematotelangiectatic Rosacea and/or Papulopustular Rosacea.
  This two arm, split-face study will consist of:
  1. Treatment arm involving treatments with 532nm KTP laser
  2. Active control arm involving treatments with 595nm Pulse Dye Laser (PDL)
  Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of treatment (532nm KTP laser) and active control treatment (595nm PDL) arms will be determined by randomization.
  Interventions: Device: 532nm KTP Laser vs 595nm Pulse Dye Laser

INTERVENTIONS:
Device: 532nm KTP Laser vs 595nm Pulse Dye Laser — Intervention for the Cutera Excel V system is to cease treatment to any subject that is experiencing any adverse reaction.

SUMMARY:
A single center prospective, randomized, controlled split face study comparing a 532nm KTP laser with a 595nm PDL for the treatment of Erythematotelangiectatic Rosacea and Papulopustular Rosacea.

Subjects will receive laser treatments and will be followed at 6 weeks post-final laser treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the 532nm KTP laser within the Cutera® Excel V system for the treatment of Erythematotelangiectatic Rosacea and Papulopustular Rosacea as compared to a 595nm Pulse Dye Laser.

The objectives of this study are:

1) To evaluate and compare the safety and efficacy of the laser treatments for Erythematotelangiectatic Rosacea and Papulopustular Rosacea at 6 weeks post final laser treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Females or Males, 20 to 80 years of age (inclusive).
2. Fitzpatrick Skin Type I - III.
3. Clinical diagnosis of Erythematotelangiectatic Rosacea and Papulopustular Rosacea.
4. Willing to refrain from using systemic corticosteroids or retinoids; or topical corticosteroids or retinoids on the treated area.
5. Must be able to read, understand and sign the Informed Consent Form.
6. Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
7. Wiling to have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the face every day for the duration of the study, including the follow-up period.
8. Willingness to have digital photographs taken of the face.
9. Agree not to undergo any other procedure for the treatment of Erythematotelangiectatic Rosacea and Papulopustular Rosacea during the study.
10. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

1. History of prior laser or light based procedures for the face within 6 months of study participation.
2. Fitzpatrick Skin Type IV - VI.
3. Pregnant and/or breastfeeding.
4. Subject is less than 20 years of age or greater than 80 years of age.
5. Having an infection, dermatitis or rash in the treatment area.
6. Suffering from significant concurrent illness, such as diabetes mellitus, cardiovascular disease, uncontrolled hypertension, or pertinent neurological disorders.
7. History of keloid formation, hypertrophic scarring or of abnormal wound healing.
8. History of immunosuppression/immune deficiency disorders such as psoriasis, eczema, vitiligo, or currently using immunosuppressive medications.
9. Malignant tumors in the target area or history of a malignant skin disease.
10. History of fibromyalgia.
11. History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
12. Having a known anticoagulative condition or taking prescription anticoagulation medications.
13. History of seizure disorders due to light.
14. Any current use of medication that is known to increase sensitivity to light, such as tetracycline.
15. Having a history of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area, unless treatment is conducted following a prophylactic regimen.
16. Having undergone any surgery in the treatment area within 6 months of treatment (or more if skin has not healed completely).
17. History of radiation to the head, neck and/or upper chest.
18. History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
19. Undergoing systemic chemotherapy for the treatment of cancer.
20. Systemic use of retinoid such as isotretinoin and/or corticosteroid within 6 months.
21. Topical use of retinoid and/or corticosteroid within 4 weeks of study participation.
22. Any use of gold therapy for disorders such as rheumatologic disease or lupus.
23. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
24. Current smoker or history of smoking within 12 months of study participation.
25. Participation in a study of another device or drug within 6 months prior to enrollment or during the study.
26. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Miami Dermatology & Laser Institute, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sides of the face
Groups:
- All Study Participants: Subjects will be treated with the Excel V 532nm (KTP) Laser and the 595nm Pulse Dye Laser: One half of the face will be treated with the 532nm KTP laser and the other half of the face will be treated with the 595nm Pulse Dye Laser.
Period: Overall Study
Arm/Group | All Study Participants
Started | 22; 44 sides of the face
Treatment With the 532nm KTP Laser | 22; 22 sides of the face
Treatment With the 595nm Pulse Dye Laser | 22; 22 sides of the face
Completed | 19; 38 sides of the face
Not Completed | 3; 6 sides of the face

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: Cutera® Excel V
  Excel V 532nm (KTP) Laser or 595nm Pulse Dye Laser: Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of treatment (532nm KTP laser) and active control treatment (595nm PDL) arms will be determined by randomization.
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Degree of Improvement in Erythematotelangiectatic Rosacea and Papulopustular Rosacea
Description: Measured for each treatment arm based on blinded physician assessment of subject photographs using the Physician's Global Assessment Scale (min=0; max=4) Higher scores mean better improvement 0 = 0% Improvement (None)
  1. = < 25% Improvement (Mild)
  2. = 26 to 50% Improvement (Moderate)
  3. = 51 to 75% Improvement (Significant)
  4. = 76 to 100% Improvement (Very Significant)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 532nm KTP Laser: Excel V 532nm (KTP) Laser on one side of the face
- 595nm Pulse Dye Laser: 595nm Pulse Dye Laser on one side of the face
Arm/Group | 532nm KTP Laser | 595nm Pulse Dye Laser
Number analyzed (Participants) | 19 | 19
score on a scale | 2.114 (1.5125) | 2.088 (1.681)

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- 532nm KTP Laser: Cutera® Excel V
  Excel V 532nm (KTP) Laser or 595nm Pulse Dye Laser: Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of treatment (532nm KTP laser) and active control treatment (595nm PDL) arms will be determined by randomization.
- 595nm Pulse Dye Laser: 595nm Pulse Dye Laser
  Excel V 532nm (KTP) Laser or 595nm Pulse Dye Laser: Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of treatment (532nm KTP laser) and active control treatment (595nm PDL) arms will be determined by randomization.
Arm/Group | 532nm KTP Laser | 595nm Pulse Dye Laser
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 22/22 | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 532nm KTP Laser (N=22) | 595nm Pulse Dye Laser (N=22)
Erythema (Skin and subcutaneous tissue disorders) | 22 | 22
Edema (Skin and subcutaneous tissue disorders) | 22 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No